CLINICAL TRIAL: NCT07006597
Title: Vitaccess Real CIDP Registry: A Prospective International Observational Patient Registry in Chronic Inflammatory Demyelinating Polyneuropathy Linking Clinical and Patient-Reported Data
Brief Title: Vitaccess Real CIDP Registry
Acronym: VRCIDP
Status: Not yet recruiting | Type: Observational
Sponsor: Vitaccess Ltd (Industry)
Responsible Party: Principal Investigator, Mark Larkin, Mark JW Larkin, PhD,Vitaccess Ltd, Vitaccess Ltd
Other Study IDs: 5166-Vitaccess-CIDP-01
Record Dates: First submitted 2025-05-27; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Chronic Inflammatory Demyelinating Polyneuropathy; CIDP
Keywords: patient registry; longitudinal observational data; patient-reported outcomes; Nervous System Disease; Autoimmune Disease; Neurodegenerative Disease; Immune System Disease; Nervous System Diseases
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating; Nervous System Diseases; Autoimmune Diseases; Neurodegenerative Diseases; Immune System Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Vitaccess Real CIDP (VRCIDP) is a patient registry designed to capture longitudinal observational data on chronic inflammatory demyelinating polyneuropathy (CIDP), its treatment, and impact on symptoms, daily activities, and quality of life (QoL). The duration of the registry is 10 years from launch, and approximately 300 patients will be recruited in the US and Europe with no defined upper limit. The registry will link relevant patient- and healthcare professional (HCP)-reported data with clinical data from electronic medical records (EMR). Patient reported and eCRF data will be linked via a unique ID and PIN assigned to each participant at enrolment.

Patients will be recruited at clinical sites in all participating countries. In the US only, patients can additionally be recruited via community neurologists or direct-to-patient recruitment.

DETAILED DESCRIPTION:
Traditional site recruitment (all countries):

Adult patients who are being treated for CIDP at one of the participating clinics or centers in one of the participating countries (the US, UK or Germany) at the time of enrolment and who meet the inclusion and exclusion criteria will be identified, approached by their clinical team and invited to participate in the registry.

Patient-reported data will be collected via the VRCIDP Registry platform, a digital data capture platform accessible via a web-enabled platform on a connected device (e.g., smartphone, tablet, laptop, computer). Custom survey and patient-reported outcomes data will be collected at baseline and at regular intervals thereafter for a follow-up period of up to 10 years. The data collected will capture the impact of CIDP on daily living, fatigue, and health-related quality of life.

Site research teams will complete and update an electronic case report form (eCRF every six months ± one month for each patient, including data from the patient's EMR. eCRFs that are completed within one months prior to or following each six-month period will be considered within the same assessment window for analytics purposes. This ensures that patients will not be required to visit the clinical site for the purposes of the registry outside of their regular clinical visits.

Community neurologist recruitment (US only):

Community neurologists who are treating CIDP patients who would be eligible for participation in the registry will be able to register their interest for involvement and provide details of their credentials via an informational website. Approved community neurologists will identify and approach potential participants, who will participate in the registry as normal. Vitaccess will partner with a third-party organization with EMR aggregator capabilities to capture data from participants' existing medical records to match eCRF outputs.

Direct-to-patient recruitment (US only):

The direct-to-patient recruitment approach will involve patients directly registering their interest for participating in the registry. Awareness of the study will be raised via collaborations with patient advisory group(s) (PAGs), who may utilize their existing relationships with CIDP patients to inform them of the study, for example via their social media. Likewise, Vitaccess may utilize social media to advertise the study directly to patients. Recruitment/promotional materials will be created for the purpose of sharing on social media platforms. As with recruitment via community neurologists, existing EMR data will be captured for consenting participants by a third-party organization with EMR aggregator capabilities.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age ≥18 years) with a clinically confirmed diagnosis of CIDP by their treating neurologist
* Resident in the US, UK or Germany
* Access to a smartphone/tablet/computer/laptop
* Willing and able to provide informed consent in their local language to take part in the study

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who are being treated for CIDP at one of the participating clinics or centers in one of the study countries (the US, UK or Germany) at the time of enrolment and who meet the inclusion and exclusion criteria will be identified and approached by their clinical team and invited to participate in the registry.
  Adult patients in the US who are not being treated at a participating clinic will be able to enrol via their community neurologist or direct-to-patient recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-07-31 (Estimated); Primary Completion 2035-07 (Estimated); Study Completion 2035-07 (Estimated)

PRIMARY OUTCOMES:
The Vitaccess Real CIDP Registry | 10 years
  A patient registry designed to build a repository of data containing disease characteristics at onset, disease progression, treatment and outcomes in CIDP [(i.e., its treatment and impact on symptoms, daily activities, and quality of life (QoL)] from patients, HCPs, and existing medical records.

SECONDARY OUTCOMES:
Describe the demographic characteristics of patients | At baseline
  EMR data reported by HCPs or captured via EMR aggregators ("Registration Form")
Describe the change in clinical trial participation of patients | At baseline visit and at follow-up visits (every 6±1 months) for up to 10 years
  EMR data reported by HCPs or captured via EMR aggregators ("Clinical Trial Participation Form")
Describe the diagnosis (date, test, symptoms) of patients | At baseline visit and at follow-up visits (every 6±1 months) for up to 10 years
  EMR data reported by HCPs or captured via EMR aggregators ("Diagnosis Information Form")
Describe the change in clinical characteristics of patients | At baseline visit and at follow-up visits (every 6±1 months) for up to 10 years
  EMR data reported by HCPs or captured via EMR aggregators ("Clinical Characteristics Form")
Describe the change in medical history of patients | At baseline visit and at follow-up visits (every 6±1 months) for up to 10 years
  EMR data reported by HCPs or captured via EMR aggregators ("Medical History Form")
Describe the change in concomitant treatments received by patients | At baseline visit and at follow-up visits (every 6±1 months) for up to 10 years
  EMR data reported by HCPs or captured via EMR aggregators ("Concomitant non-CIDP medications log")
Describe the change in routine CIDP treatments received by patients | At baseline visit and at follow-up visits (every 6±1 months) for up to 10 years
  EMR data reported by HCPs or captured via EMR aggregators ("Routine CIDP medication log")
Describe change in rescue CIDP treatments received by patients | At baseline visit and at follow-up visits (every 6±1 months) for up to 10 years
  EMR data reported by HCPs or captured via EMR aggregators ("Rescue CIDP Treatments Log")
Describe the change in healthcare resource use of patients | At baseline visit and at follow-up visits (every 6±1 months) for up to 10 years
  EMR data reported by HCPs or captured via EMR aggregators ("Healthcare Resource Use")
Describe change in type and severity of adverse events experienced by patients | At baseline visit and at follow-up visits (every 6±1 months) for up to 10 years
  EMR data reported by HCPs or captured via EMR aggregators ("Adverse Events Form")
Describe change in caregiver requirements experienced by patients | At baseline visit and at follow-up visits (every 6±1 months) for up to 10 years
  EMR data reported by HCPs or captured via EMR aggregators ("Caregiver Information Form")
Describe the family history of patients | At baseline visit and at follow-up visits (every 6±1 months) for up to 10 years
  EMR data reported by HCPs or captured via EMR aggregators ("Family History Form")
Describe the change in employment status of patients | At baseline visit and at follow-up visits (every 6±1 months) for up to 10 years
  EMR data reported by HCPs or captured via EMR aggregators ("Employment Status Form")
Describe the change in health insurance status and out-of-pocket costs experienced by patients | At baseline visit and at follow-up visits (every 6±1 months) for up to 10 years
  EMR data reported by HCPs or captured via EMR aggregators ("Health Insurance Status Form")
Describe the disease history of patients | At baseline visit and at follow-up visits (every 6±1 months) for up to 10 years
  EMR data reported by HCPs or captured via EMR aggregators ("Disease History")
Describe the clinical investigations performed by treating neurologists on patients | At baseline visit and at follow-up visits (every 6±1 months) for up to 10 years
  EMR data reported by HCPs or captured via EMR aggregators ("Clinical Investigations")
Describe the treatment decisions and rationale for treatment decisions made by treating neurologists | At baseline visit and at follow-up visits (every 6±1 months) for up to 10 years
  EMR data reported by HCPs or captured via EMR aggregators ("Management Decisions by Treating Neurologist", "Health System Implications on Treatment", "Patient Choice on Treatment Decisions", "Tools used for Therapeutic Decisions")
Describe the impact of CIDP on multiple life domains | At baseline and every 6 months thereafter for up to 10 years.
  "Chronic Acquired Polyneuropathy patient-reported index (CAP-PRI)" data reported by patients via the Vitaccess Real CIDP Registry platform
Describe the impact of CIDP on work productivity and daily activities | At baseline and every 6 months thereafter for up to 10 years.
  "Work Productivity and Activity Impairment (WPAI)" data reported by patients via the Vitaccess Real CIDP Registry platform
Describe the health-related quality of life (HRQoL) of patients | At baseline visit and every 3 months thereafter for up to 10 years.
  "EQ-5D-5-level version (EQ-5D-5L)" data reported by patients via the Vitaccess Real CIDP Registry platform
Describe the fatigue levels of patients | At baseline visit and every 6 months thereafter for up to 10 years.
  "NeuroQoL Fatigue Short Form" data reported by patients via the Vitaccess Real CIDP Registry platform
Describe the stress levels of patients | At baseline visit and every 6 months thereafter for up to 10 years.
  "Perceived Stress Fixed Form" data reported by patients via the Vitaccess Real CIDP Registry platform
Describe the pain of patients | At baseline visit and every 6 months thereafter for up to 10 years.
  "PROMIS Neuropathic Pain Quality 5a" and "PROMIS Pain Intensity 3a" data reported by patients via the Vitaccess Real CIDP Registry platform
Describe the impact of CIDP on mood | At baseline visit and every 6 months thereafter for up to 10 years.
  "Hospital Anxiety and Depression Scale (HADS)" data reported by patients via the Vitaccess Real CIDP Registry platform
Describe the perceived change in CIDP since study start | At baseline visit and every 6 months thereafter for up to 10 years.
  "Patient global impression of change (PGIC)" data reported by patients via the Vitaccess Real CIDP Registry platform

IPD SHARING:
Plan to Share IPD: No